CLINICAL TRIAL: NCT00773864
Title: Mastering Hospital Antimicrobial Resistance and Its Spread Into the Community- the Role of Healthcare Workers
Brief Title: Mastering Hospital Antimicrobial Resistance and Its Spread Into the Community-Healthcare Workers
Acronym: MOSAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: yaffa lerman, MD, TASMC
Other Study IDs: TASMC-08-YC-254-CTIL
Record Dates: First submitted 2008-10-06; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus; ESBL
Keywords: Healthcare employees who work in the rehabilitation center

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Medical staff will be screened for MRSA and ESBL (including: doctors, nurses, nurse aids, physical therapists, dietitians, Janitors and other medical staff).

PURPOSE:

To define the carriage of, and risk factors for carriage of resistant organisms among healthcare employees of carriers of resistant bacteria.

To define activities of healthcare employees who likely to lead to dissemination of resistant bacteria in rehabilitation centers.

DETAILED DESCRIPTION:
Detailed activity:

Medical staff will be screened for MRSA and ESBL (including: doctors, nurses, nurse aids, physical therapists, dietitians, Janitors and other medical staff).

Screening will be performed by obtaining nares and perirectal cultures. Nares cultures will be obtained by ward staff or research personnel who are experienced in performing this activity: a moisture swab will be applied gently to the distal part of both nares. Perirectal cultures, will be taken by swab, who will be applied to the perirectal area, either by staff as mentioned above, or will be given to the healthcare workers to perform by himself (with explanation on how to perform it).

ELIGIBILITY:
Inclusion Criteria:

* Health care employees

Exclusion Criteria:

* Age 18 years or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare employees) including: doctors, nurses, nurse aids, physical therapists, dietitians, Janitors and other medical staff) who work in the rehabilitation center
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Healthcare employees) including: doctors, nurses, nurse aids, physical therapists, dietitians, Janitors and other medical staff) who work in the rehabilitation center | 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda carmeli, MD MPH, Principal Investigator — TASMC
Locations (1):
- Tasmc, Tel Aviv, Israel

REFERENCES:
- [Background] Albrich WC, Harbarth S. Health-care workers: source, vector, or victim of MRSA? Lancet Infect Dis. 2008 May;8(5):289-301. doi: 10.1016/S1473-3099(08)70097-5. PMID 18471774
- [Background] Carmeli Y, Venkataraman L, DeGirolami PC, Lichtenberg DA, Karchmer AW, Samore MH. Stool colonization of healthcare workers with selected resistant bacteria. Infect Control Hosp Epidemiol. 1998 Jan;19(1):38-40. doi: 10.1086/647705. PMID 9475348